CLINICAL TRIAL: NCT03366103
Title: Phase 1/2 Study of Navitoclax Plus Vistusertib in Patients With Relapsed Small Cell Lung Cancer (SCLC) and Other Solid Tumors
Brief Title: Navitoclax and Vistusertib in Treating Patients With Relapsed Small Cell Lung Cancer and Other Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00037; NCI-2017-00037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ETCTN10070; 10070 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10070 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2017-12-07; First posted 2017-12-08 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Malignant Solid Neoplasm; Recurrent Lung Small Cell Carcinoma; Recurrent Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Stage III Lung Small Cell Carcinoma, by American Joint Committee on Cancer (AJCC) v7; Stage IIIA Lung Small Cell Carcinoma AJCC v7; Stage IIIB Lung Small Cell Carcinoma AJCC v7; Stage IV Lung Small Cell Carcinoma AJCC v7; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Small Cell Lung Carcinoma | interventions — navitoclax; vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (navitoclax, vistusertib) (Experimental): Patients receive navitoclax PO QD and vistusertib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Navitoclax; Drug: Vistusertib

INTERVENTIONS:
Biological: Navitoclax — Given PO
  Other Names: A-855071.0; ABT-263; BcI-2 Family Protein Inhibitor ABT-263
Drug: Vistusertib — Given PO
  Other Names: AZD 2014; AZD-2014; AZD2014

SUMMARY:
This phase I/II trial studies the best dose and side effects of navitoclax and how well it works when given together with vistusertib in treating patients with small cell lung cancer and solid tumors that have come back (relapsed). Drugs used in chemotherapy, such as navitoclax, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Vistusertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving navitoclax and vistusertib may work better than navitoclax alone in treating patients with small cell lung cancer and solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of navitoclax and vistusertib in patients with advanced solid tumors. (Phase I) II. To determine the maximum tolerated dose (MTD), dose limiting toxicities (DLT), and recommended phase 2 doses (RP2D) of navitoclax and vistusertib. (Phase I) III. To determine the objective response rate (ORR), defined as complete plus partial response, of the combination of navitoclax and vistusertib in patients with recurrent small cell lung cancer (SCLC). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of navitoclax and vistusertib when administered together. (Phase I) II. To observe and record anti-tumor activity. (Phase I) III. To confirm the safety and tolerability of navitoclax and vistusertib at the RP2D. (Phase II) IV. To estimate progression free survival (PFS) and overall survival (OS) of the combination of navitoclax and vistusertib at the RP2D. (Phase II) V. To estimate disease control rate (DCR) of the combination of navitoclax and vistusertib at the RP2D. (Phase II)

CORRELATIVE OBJECTIVES:

I. To assess pharmacodynamic changes in levels of phosphorylated 4EBP1 (p4EBP1) the ratio of p4EBP1 to total (p4EBP1/4EBP1) in paired pre-treatment and on-treatment biopsies at the RP2D. (Phase II) II. To correlate changes in BAX and MCL-1 with response. (Phase II) III. To estimate the baseline inter-patient variability in p4EBP1, pS6, BAX, and MCL-1. (Phase II) IV. To explore exposure-response relationships between navitoclax and vistusertib exposure and the pharmacodynamic endpoints (safety, efficacy, and laboratory correlatives). (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive navitoclax orally (PO) once daily (QD) and vistusertib PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 8-12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE 1 SPECIFIC ELIGIBILITY CRITERIA
* Patients must have histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* PHASE 2 SPECIFIC ELIGIBILITY CRITERIA
* Patients must have histologically or cytologically confirmed small cell lung cancer whose disease has relapsed or progressed after >= 1 prior therapy, one of which must have been a platinum doublet; pathology confirmation must be done at Sidney Kimmel Comprehensive Cancer Center (SKCCC) or at the local participating site
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Subjects must be willing to undergo 2 sets of core needle biopsies (pre-treatment and on-treatment), if there are lesions amenable to biopsy; an optional core biopsy will be requested at progression
* GENERAL ELIGIBILITY CRITERIA
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9.0 g/dL
* Platelets >= 100,000/mcL
* Activated partial thromboplastin time (aPTT), prothrombin time (PT) =< 1.2 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN (patients with Gilbert's syndrome may have serum bilirubin > 1.5 ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN if no demonstrable liver metastases or =< 5 x ULN in the presence of liver metastases
* Creatinine =< 1.5 x ULN and concurrent creatinine clearance (CrCl) >= 50 mL/min/1.73 m^2 for patients with creatinine (Cr) > 1.5 x ULN
* Proteinuria < 1+ on dipstick testing (if 2+ seen on first test, retest >= 24 hours later)
* Patients with a history of central nervous system (CNS) metastases must have documentation of stable or improved status based on brain imaging for at least 2 weeks after completion of definitive treatment and within 2 weeks prior to first dose of study drug, off or on a stable dose of corticosteroids
* Patients must have completed chemotherapy, biological or radiotherapy >= 3 weeks prior to entering the study
* Patients must have recovered to =< grade 1 adverse events or to =< grade 2 alopecia and sensory neuropathy due to prior treatment
* Patients must be able to understand and the willingness to sign a written informed consent document
* Patients must be able to swallow pills
* The effects of navitoclax and vistusertib on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and up to 90 days following completion of therapy; for women this should include one highly effective method of contraception and one barrier method as defined below

  * Highly effective methods include:

    * Total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to study drug administration);
    * Vasectomized partner;
    * Medroxyprogesterone acetate depot injection;
    * Placement of a copper-banded intrauterine device (IUD) or intrauterine system (IUS);
    * Bilateral tubal ligation;
  * Barrier methods include:

    * Condom;
    * Occlusive cap (e.g. diaphragm or cervical/vault caps) with spermicide
  * Please note: use of other oral, injected or implanted hormonal methods of contraception cannot be considered highly effective as it is currently unknown whether vistusertib may reduce their effectiveness; periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception
  * Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 90 days following completion of therapy
* Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to initiation of treatment, women will be considered not of childbearing potential if they are surgically sterile (bilateral oophorectomy or hysterectomy) and/or post-menopausal (amenorrheic for at least 12 months)
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 90 days after completion of navitoclax and/or vistusertib administration

Exclusion Criteria:

* PHASE 2 SPECIFIC EXCLUSION CRITERIA
* Prior treatment with a TORC1, dual TORC1/2 inhibitor, or BCL-2/xL inhibitor
* Patients with active malignancies other than SCLC or patients with prior curatively treated malignancy at high risk of relapse during the study period with the exception of localized squamous or basal cell skin cancers
* PHASE 1 AND GENERAL EXCLUSION CRITERIA
* Major surgery within 21 days of starting protocol treatment
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to navitoclax or vistusertib
* Patients receiving anticoagulation or anti-platelet therapy are excluded due to the risk of thrombocytopenia with navitoclax

  * Excluded agents include heparin or low molecular weight heparin, warfarin, clopidogrel, ibuprofen and other non-steroidal anti-inflammatory drugs (NSAIDS), tirofiban, and other anticoagulants, drugs, or herbal supplements that affect platelet function
  * Administration of heparin to keep subject's infusion lines patent is allowed; low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter are allowed
  * Aspirin will not be allowed within 7 days prior to the first dose of navitoclax or during navitoclax administration; however, subjects who have previously received aspirin therapy for thrombosis prevention, may resume a low dose (i.e., maximum 100 mg once daily [QD]) of aspirin if platelet counts are stable (>= 50,000/mm3) through 6 weeks of navitoclax administration
  * All decisions regarding treatment with aspirin therapy will be determined by the investigator in conjunction with the medical monitor
* Patients with an underlying condition predisposing them to bleeding or currently exhibiting signs of clinically significant bleeding
* Patients with a recent history of non-chemotherapy-induced thrombocytopenic-associated bleeding within 1 year prior to the first dose of study drug
* Patients with a significant history of cardiovascular disease or procedures within the preceding 6 months (e.g., myocardial infarction [MI], coronary artery bypass graft placement, angioplasty, vascular stent, angina pectoris, ventricular arrhythmias requiring continuous therapy, congestive heart failure New York Heart Association [NYHA] grade >= 2, thrombotic or thromboembolic event)
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc using Fridericia's formula [QTcF]) > 470 msec obtained from 3 electrocardiograms
  * Congenital or family history of long or short QT syndrome, Brugada syndrome, known history of QTc prolongation or torsades de pointes within 12 months of entering the study
  * Abnormal echocardiogram at baseline (left ventricular ejection fraction [LVEF] < 40% and shortening fraction [SF] < 15%)
* Drugs which have an increased risk for QTc prolongation should be avoided
* Patients with uncontrolled type 1 or type 2 diabetes. Vistusertib belongs to a class of drugs that causes hyperglycemia. In order to assess toxicity, patients with an elevated risk of hyperglycemia should be excluded from study
* Patients currently receiving medications or herbal supplements of the classes below are ineligible; patients are eligible if they stop use of these compounds at least 1 week prior to receiving any treatment on this protocol

  * Potent inhibitors or inducers of CYP3A4 /5 (CYP3A4 inhibitors such as ketoconazole and clarithromycin are not allowed 7 days prior to the first dose of navitoclax and during navitoclax administration)
  * Strong or moderate inhibitors of Pgp or BRCP1
  * Sensitive substrates of CYP2C9 (i.e. phenytoin and warfarin)
  * Substrates of certain drug transporters (OATP1B1, OATP1B3, MATE1 or MATE2K)
* Pregnant women are excluded from this study because navitoclax and vistusertib have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with navitoclax and vistusertib breastfeeding should be discontinued if the mother is treated with navitoclax and vistusertib
* Patients positive for human immunodeficiency virus (HIV) are not excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART) that does not include strong or moderate CYP3A4 inducers or inhibitors
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based test
* Any hematopoietic growth factors (e.g., filgrastim [granulocyte colony-stimulating factor; G-CSF], sargramostim [granulocyte-macrophage colony-stimulating factor; GM-CSF]) within 14 days prior to receiving study treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have received a live, attenuated vaccines within 4 weeks of first dose of drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine L Hann, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (14):
- United States (14):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Scott SC, Farago A, Lai WV, Zahurak M, Rudek MA, Murray J, Carducci MA, Uziel T, Takebe N, Gore SD, Rudin CM, Hann CL. A phase 1 study of the combination of BH3-mimetic, navitoclax, and mTORC1/2 inhibitor, vistusertib, in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2025 Feb 25;95(1):37. doi: 10.1007/s00280-025-04760-1. PMID 39998620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1: 03/20/2018 - 11/11/2019 Phase 2: 7/29/2020 - 5/19/2021
Groups:
- Phase 1 - Dose Level 1; Phase 2: Navitoclax 150 mg po qd + Vistusertib 35 mg po bid
- Phase 1 - Dose Level 2: Navitoclax 250 mg po qd + Vistusertib 35 mg po bid
Period: Overall Study
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2
Started | 9 | 5 | 1
Completed | 6 | 3 | 1
Not Completed | 3 | 2 | 0
Not completed — Disease Progression | 3 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 - Dose Level 1: Patients receive navitoclax 150 mg orally (PO) once a day (QD) and vistusertib 35 mg PO twice a day (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 - Dose Level 2; Phase 2: Patients receive navitoclax 250 mg PO QD and vistusertib 35 mg PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2 | Total
Number analyzed (Participants) | 9 | 5 | 1 | 15
Age, Continuous [Median (Full Range); unit: years] | 49 [35 to 74] | 67 [53 to 71] | 77 [77 to 77] | 60 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 0 | 9
  Male | 3 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 1 | 14
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 7 | 4 | 1 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 1 | 15
Weight [Median (Full Range); unit: kg] | 75 [58.5 to 86.8] | 68.5 [56.6 to 114.4] | 86.2 [86.2 to 86.2] | 75 [56.6 to 114.4]
Height [Median (Full Range); unit: cm] | 167.6 [162.6 to 188.0] | 165.0 [162.5 to 178.0] | 172.7 [172.7 to 172.7] | 167.6 [162.5 to 188]
Body Surface Area (BSA) [Median (Full Range); unit: m^2] | 1.90 [1.63 to 2.00] | 1.76 [1.62 to 2.31] | 2.03 [2.03 to 2.03] | 1.9 [1.62 to 2.31]
Primary site of disease [Count of Participants; unit: Participants]
  Appendix | 1 | 0 | 0 | 1
  Breast | 2 | 0 | 0 | 2
  Cervix | 1 | 0 | 0 | 1
  Colon | 2 | 0 | 0 | 2
  Lung | 2 | 5 | 1 | 8
  Pleura | 1 | 0 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  Asymptomatic | 2 | 1 | 0 | 3
  Symptomatic, fully ambulatory | 7 | 3 | 1 | 11
  Able to carry on normal activity, minor symptoms | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (Phase I)
Description: Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0. The number of participants with dose limiting toxicities at each dose level will be reported with exact binomial 95% confidence intervals. All patients who receive at least 1 dose of both study drugs, regardless of their eligibility for the study, will be evaluable for toxicity.
Time Frame: Up to 30 days after last treatment, an average of 3 months
Population: Phase 1 participants were included in this analysis. Please see AE section for additional details.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2
Number analyzed (Participants) | 6 | 3
Participants
  DLT | 0 | 2
  No DLT | 6 | 1

2. Primary Outcome: Overall Response Rate (ORR) (Phase II)
Description: Defined as Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. partial response or complete response, of the combination in patients with recurrent small cell lung cancer. The ORR will be reported with its corresponding 95% confidence interval.
Time Frame: Up to 1.5 years
Population: Only one participant was enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 1
Participants
  Partial Response (PR) or Complete Response (CR) | 0
  Stable Disease (SD) | 0
  Progression (PD) | 1

3. Secondary Outcome: Occurrence of a Bi-directional Pharmacokinetic (PK) Interaction
Description: Concentrations of each study agent present in the blood at the specified time point are reported for each study agent.
Time Frame: Through Day 15
Population: Participants in both phases were included. Some data was not collected at each timepoint.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Navitoclax 150 mg + Vistusertib 35 mg: Participants in either Phase who received Navitoclax 150 mg.
- Navitoclax 250 mg + Vistusertib 35 mg: Participants in either Phase who received Navitoclax 250 mg
- Navitoclax 250 mg Reduced to 150 mg + Vistusertib 35 mg: Participants who initially received Navitoclax 250 mg but were reduced to navitoclax 150 mg.
Arm/Group | Navitoclax 150 mg + Vistusertib 35 mg | Navitoclax 250 mg + Vistusertib 35 mg | Navitoclax 250 mg Reduced to 150 mg + Vistusertib 35 mg
Number analyzed (Participants) | 9 | 5 | 1
ng/ml
  Navitoclax average of individual steady-state trough concentration (avg Cmin,ss) | 1145 (289) | 1966 (999) | 2283
  Navitoclax Cycle 1 Day 1 Concentration 6 hours after dose (C6h): number analyzed (Participants) | 4 | 5 | 0
  Navitoclax Cycle 1 Day 1 Concentration 6 hours after dose (C6h) | 1808 (980) | 3254 (1233) |
  Navitoclax Cycle 1 Day 15 Concentration 6 hours after dose (C6h): number analyzed (Participants) | 6 | 2 | 1
  Navitoclax Cycle 1 Day 15 Concentration 6 hours after dose (C6h) | 2260 (993) | 2830 (1190) | 3450
  Navitoclax Cycle 1 Day 15 maximum concentration (Cmax): number analyzed (Participants) | 6 | 2 | 1
  Navitoclax Cycle 1 Day 15 maximum concentration (Cmax) | 2393 (913) | 3060 (1070) | 3910
  Vistusertib average of individual steady-state trough concentration (avg Cmin,ss): number analyzed (Participants) | 9 | 4 | 1
  Vistusertib average of individual steady-state trough concentration (avg Cmin,ss) | 211 (207) | 559 (550) | 238.5
  Vistusertib Cycle 1 Day 1 Concentration 2 hours after dose (C2h): number analyzed (Participants) | 4 | 5 | 0
  Vistusertib Cycle 1 Day 1 Concentration 2 hours after dose (C2h) | 372 (266) | 419 (108) |
  Vistusertib Cycle 1 Day 15 Concentration 2 hours after dose (C2h): number analyzed (Participants) | 6 | 3 | 1
  Vistusertib Cycle 1 Day 15 Concentration 2 hours after dose (C2h) | 1061 (675) | 1032 (832) | 273

4. Secondary Outcome: Number of Participants Experiencing Adverse Events by Grade (Phase II)
Description: Graded by NCI CTCAE v 4.0. The number of participants with toxicities by grade in the phase 2 study will be reported with exact binomial 95% confidence intervals.
Time Frame: Up to 1.5 years
Population: Only one participant was enrolled.
Measure: Number; unit: participants
Arm/Group | Phase 2
Number analyzed (Participants) | 1
participants
  Grade 1 Adverse Events | 1
  Grade 2 Adverse Events | 1
  Grade 3 Adverse Events | 0
  Grade 4 Adverse Events | 0
  Grade 5 Adverse Events | 0

5. Secondary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Based on RECIST 1.1. Standard life table methods will be used to analyze PFS. We will report the one-year and median PFS with 95% confidence intervals.
Time Frame: Up to 1.5 years
Population: Only one participant was enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Overall Survival (OS) at Year 1 (Phase II)
Description: Standard life table methods will be used to analyze OS. We will report the one-year and median OS with 95% confidence intervals.
Time Frame: At Year 1
Population: Only one participant was enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Disease Control Rate (Phase II)
Description: Based on RECIST 1.1. The proportion of patients achieving disease control will be reported with exact 95% binomial confidence intervals.
Time Frame: Up to 1.5 years
Population: Only one participant was enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 1
Participants | 0

8. Other Pre Specified Outcome: Change in p4EBP1 Expression
Description: Descriptive statistics and box plots with jittered data points will be used to visualize all raw data. Will be assessed with paired t-tests.
Time Frame: Baseline up to 1.5 years
Population: Data was not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Change in Ratio p4EBP1/4EBP1
Description: as for outcome 8
Time Frame: Baseline up to 1.5 years
Population: Data was not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Change in Ratio pS6/S6
Description: as for outcome 8
Time Frame: Baseline up to 1.5 years
Population: Data was not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Change in BAX and MCl-1 Expression
Description: as for outcome 8
Time Frame: Baseline up to 1.5 years
Population: Data was not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Pharmacodynamic Parameters
Description: Exploratory correlative studies with pharmacodynamic (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics.
Time Frame: Up to 1.5 years
Population: Data was not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1.5 years
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 6/9 | 3/5 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose Level 1 (N=9) | Phase 1 - Dose Level 2 (N=5) | Phase 2 (N=1)
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Blood bilirubin decreased (Investigations) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose Level 1 (N=9) | Phase 1 - Dose Level 2 (N=5) | Phase 2 (N=1)
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Cramping (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Frequent stool (Gastrointestinal disorders) | 1 | 0 | 0
Loose stool (Gastrointestinal disorders) | 1 | 0 | 0
Thrush (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 0
Edema limbs (General disorders) | 0 | 1 | 0
Fever (General disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Sweating (General disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0
Weight loss (Investigations) | 0 | 2 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
INR increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cramping (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Renal and urinary disorders (Renal and urinary disorders) | 0 | 0 | 1 — Urinary burning
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — Hypersensitivity
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Death NOS (General disorders) | 2 | 1 | 0
Progressive Disease (General disorders) | 3 | 2 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Only 1 participant was enrolled to Phase 2 before the study was closed to accrual for low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03366103/Prot_SAP_000.pdf